CLINICAL TRIAL: NCT05446558
Title: Long-term Clinical Results and Direct Economic Implication Within the Randomized Clinical Trial Comparing Intracorporeal Versus Extracorporeal Anastomosis in Laparoscopic Right Colectomy
Brief Title: Long-term Results in Intracorporeal Versus Extracorporeal Anastomosis in Laparoscopic Right Colectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-ANA-2021-16
Record Dates: First submitted 2022-05-23; First posted 2022-07-06 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Colon Cancer; Colon Neoplasm; Malignant Neoplasm; Colon Neoplasia; Colon Neoplasm, Malignant
Keywords: anastomosis; laparoscopic right colectomy; intracorporeal; extracorporeal; intracorporeal anastomosis; extracorporeal anastomosis; randomized controlled trial; oncological outcomes; long-term follow-up; colectomy; minimally invasive surgery
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: The study was a parallel group trial with a 1:1 allocation ratio.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracorporeal anastomosis (IA) (Experimental): Experimental: Intracorporeal anastomosis Iso or anti-peristaltic side-to-side ileo-colonic anastomosis with Echelon Endopatch and closure of the defect with running suture or another firing of Echelon Endopatch. The surgical specimen is retrieved through a Pfannenstiel incision.
  Interventions: Procedure: Intracorporeal anastomosis
- Extracorporeal anastomosis (EA) (Active Comparator): A transverse incision in the right upper quadrant is performed. An iso or anti-peristaltic side-to-side ileo-colonic anastomosis with Proximate Linear Cutter device and Proximate Rel Stapler
  Interventions: Procedure: Extracorporeal anastomosis

INTERVENTIONS:
Procedure: Intracorporeal anastomosis — Iso or anti-peristaltic side-to-side ileo-colonic anastomosis with Echelon Endopatch and closure of the defect with running suture or another firing of Echelon Endopatch. The surgical specimen will be retrieved through a Pfannenstiel incision.
  Device:
  Use of an Echelon Endopatch Powered Device to perform an ileocolonic side-to-side anastomosis.
  Arms: Intracorporeal anastomosis (IA)
Procedure: Extracorporeal anastomosis — A transverse incision in the right upper quadrant will be performed. An iso or anti-peristaltic side-to-side ileo-colonic anastomosis with Proximate Linear Cutter device and Proximate Stapler.
  Device:
  Use of a Proximate Linear Cutter device to perform a side-to-side ileo-colonic anastomosis.Use of a Proximate stapler to the closure of the defect associated with the creation of the side-to-side ileo-colonic anastomosis.
  Arms: Extracorporeal anastomosis (EA)

SUMMARY:
Advantages of laparoscopic right colectomy with intracorporeal anastomosis (IA) compared to extracorporeal anastomosis (EA) are widely studied. Nowadays we can conclude, with a high level of scientific evidence, that there are a number of short-term clinical advantages of laparoscopic right colectomy with intracorporeal anastomosis (IA).

However, there is currently no randomized studies describing long-term clinical and oncological outcomes.

DETAILED DESCRIPTION:
Background:

Little evidence has been published demonstrating the advantages of IA versus EA.

Recent publications show the superiority of IA in terms of early functional digestive recovery, a shorter surgical incision, a lower need for analgesia, lower blood loss, and lower postoperative Clavien-Dindo grade. These results are similar to other further published studies, including multicenter randomized clinical trials and meta-analyses.

Methods:

This is a a long-term clinical follow-up study of 140 patients included preaviously in the single-blind single-center randomized prospective clinical trial conducted at the Hospital de la Santa Creu i Sant Pau (HSCSP) between 2015-2018; in which 30-day clinical outcomes after laparoscopic right colectomy for colon cancer with IA vs EA anastomosis were compared.

In this new trial, prospective clinical follow-up of the included 140 patients, randomized in two groups IA and EA, will be carried out, with a minimum time of 3 years.

The main objective of the study will be:

-Comparing long-term oncological outcomes of IA vs. EA anastomosis in laparoscopic right colectomy for malignant neoplasm.

The secondary objectives will be:

* Analyzing the appearance of abdominal wall hernias and episodes of occlusion.
* Describing the direct costs of both techniques retrospectively, through the financial records of the HSCSP institution.

The main hypothesis will be:

-IA is not inferior compared to EA in terms of oncological and clinical results, with a lower rate of abdominal postoperative hernias and occlusive/subocclusive episodes.

A regular prospective clinical follow-up through periodic medical visits and complementary tests established by the criteria of the Colorectal Cancer management protocol (document agreed by the HSCSP Colorectal Tumors Committee) will be conducted.

For the economic evaluation, all direct in-hospital costs that were registered by the HSCSP management will be analysed.

Extensive written information and an informed consent about the study will be provided to the patient.

The study does not entail any risk for the patient as it does not interfere with the usual follow-up or require extraordinary complementary studies.

ELIGIBILITY:
Inclusion Criteria:

* Neoplasms settled in the cecum, right colon, hepatic flexure or proximal transverse colon
* Surgical procedure with curative purpose.
* American Society of Anaesthesiologists Physical Status (ASA) I, II and III.
* Elective surgery.
* Signed Informed Consent.

Exclusion Criteria:

* Denial of informed consent.
* Advanced neoplasia (Stage IV)
* Urgent surgery.
* ASA IV.
* Bening colonic disease, such Ulcerative Colitis or Crohn Disease
* Multivisceral procedures performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-28 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Percentage of patients alive after a 3-years follow-up-period since the laparoscopic right colectomy is performed

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  Percentage of patients alive without any type of recurrence (local or distant) after a 3-years follow-up-period since the laparoscopic right colectomy is performed
Local recurrence | 3 years
  Percentage of patients that experiment disease recurrence which is placed in the previously operated area
Distant recurrence | 3 years
  Percentage of patients that experiment disease recurrence which is placed in a different area from the previously operated region (intraperitoneal, liver, lung metastases, etc)
Incisional hernia | 3 years
  Percentage of patients that present an abdominal hernia settled on any of the incisions performed during the laparoscopic right colectomy
Intestinal obstruction | 3 years
  Percentage of patients that experiment mechanical impairment or complete arrest of the passage of contents through the intestine due to pathology that causes blockage of the bowel.
Cost of surgical material | Intraoperative time
  Price (in euro) of the material used in the operating room in each procedure
Cost of operative room | Intraoperative time
  Price (in euro) of the total amount of hours of surgical time per each procedure
Cost per global hospitalization | Time from the first day of operation until the day that the patient is discharged from the hospital
  Price (in euro) of the total amount of days of hospitalization per each group
Cost per ICU hospitalization | Time from the first day of entry into ICU until the day that the patient is transfered to Surgery Department
  Price (in euro) of the total amount of days of hospitalization in Intensive Care Unit per each group
Cost of tests during hospitalization | Time from the first day of operation until the day that the patient is discharged from the hospital
  Price (in euro) of the total amount of costs related to laboratory and diagnosis during the hospitalization period, per each group

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Background] Bollo J, Salas P, Martinez MC, Hernandez P, Rabal A, Carrillo E, Targarona E. Intracorporeal versus extracorporeal anastomosis in right hemicolectomy assisted by laparoscopy: study protocol for a randomized controlled trial. Int J Colorectal Dis. 2018 Nov;33(11):1635-1641. doi: 10.1007/s00384-018-3157-9. Epub 2018 Sep 6. PMID 30191370
- [Background] Bollo J, Turrado V, Rabal A, Carrillo E, Gich I, Martinez MC, Hernandez P, Targarona E. Randomized clinical trial of intracorporeal versus extracorporeal anastomosis in laparoscopic right colectomy (IEA trial). Br J Surg. 2020 Mar;107(4):364-372. doi: 10.1002/bjs.11389. Epub 2019 Dec 17. PMID 31846067